CLINICAL TRIAL: NCT06234319
Title: Clinical Study on CXCR4 PET/MRI Targeted Integrated Imaging for Grading Diagnosis, Molecular Typing, and Prognostic Evaluation of Brain Glioma
Brief Title: CXCR4 PET/MRI Targeted Imaging for Grading Diagnosis, Molecular Typing, and Prognostic Evaluation of Brain Glioma
Status: Recruiting | Type: Observational
Sponsor: Xiao Chen (Other)
Responsible Party: Sponsor-Investigator, Xiao Chen, Director of Nuclear Medicine Department, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Other Study IDs: 20230294
Record Dates: First submitted 2024-01-04; First posted 2024-01-31 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — brain glioma resction specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CXCR4 — Patients with clinical suspected primary glioma will receive a CXCR4 PET imaging.

SUMMARY:
This project intends to evaluate the role of C-X-C chemokine receptor type 4 (CXCR4) targeted PET/MRI integrated imaging in the grading and molecular typing of brain gliomas, using primary glioma patients as the research subjects and post-operative histopathological analysis as the reference, and to establish an evaluation model for the prognosis of primary glioma patients.

DETAILED DESCRIPTION:
1. PET/MRI Scan: Image acquisition was completed 15 days before surgery. CXCR4 contrast agent was injected at 6.5 MBq/kg based on body mass, with no drug extravasation, and imaging was performed after 60 minutes of quiet rest. All subjects were scanned in a supine position on a single bed of the Signa™ 3.0T scanner (GE Healthcare Systems), using a 3.0T gem HNU head coil with a scanning field of view focused on the head. PET acquisition lasted for 20 minutes and was reconstructed using OSEM. Simultaneous MRI acquisition included MR-based attenuation correction (MRAC) - zero echo time pulse sequence (ZTE), as well as structural and functional MRI sequences (T1WI, T2WI, FLAIR, DWI, MRS, DSC, T1-CE). Image fusion was performed on a GE post-processing workstation.
2. Image Analysis and Observation Indicators: PET/MRI images were independently reviewed and processed by two experienced neuroradiologists. Using IKT-SNAP software, target lesion VOIs were outlined based on FLAIR and T1-CE sequences. VOI delineation on the FLAIR sequence included solid tumor components, necrotic areas, and surrounding abnormal FLAIR signal regions. VOI delineation on the T1-CE sequence included enhanced solid components, non-enhanced solid components, and necrotic areas. MRI parameters (diffusion-weighted imaging parameters: ADC; perfusion imaging parameters: CBF, CBV, MTT, TTP; spectroscopic parameters: NAA, Cho, Cr, Lac, NAA/Cr, Cho/Cr) and PET parameters (SUVmax, SUVmean, SUVpeak, CXCR4 metabolic volume, TBR) were measured throughout the tumor and corresponding regions.
3. Pathological Analysis: Slices containing no less than 25% tumor tissue were used, with each slice having a thickness of 4um. HE, CD34, and CXCR4 immunohistochemical staining were performed separately. Two senior pathologists reviewed the slides using a double-blind method. IDH mutation status and 1p/19q deletion status were determined by the pathology department.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with primary glioma based on clinical, imaging, and histopathological criteria;
2. The patient is at least 18 years old;
3. Participate in CXCR4 PET/MRI imaging within 15 days before surgery;
4. Surgical resection of glioma lesion tissue can be used for pathological analysis;
5. The patient voluntarily participates and signs the informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding patients;
2. The image quality of the imaging is poor and cannot be used for diagnosis and evaluation;
3. Molecular typing was not determined by histologic examination;
4. patients with claustrophobia;
5. Patients who are allergic to radioactive tracers and MRI contrast agents, and patients with renal insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects are adults with newly diagnosed primary glioma, regardless of gender.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardised uptake values | completed within one week after the PET/MRI examination
  Standardised uptake values of suspected glioma disease in CXCR4 PET/MRI imaging
expression of CD34 | completed within one week after surgery
  Immunohistochemical evaluation of the expression of CD34 in postoperative tumor tissue
expression of CXCR4 | completed within one week after surgery
  Immunohistochemical evaluation of the expression of CXCR4 in postoperative tumor tissue

SECONDARY OUTCOMES:
SUV and histological grading of glioma | through study completion, an average of 1 year
  Correlation between SUV and histological grading of glioma
CXCR4 expression and histological grading of glioma | through study completion, an average of 1 year
  Correlation between CXCR4 expression and histological grading of glioma
SUV and IDH mutation status | through study completion, an average of 1 year
  Correlation between SUV and IDH mutation status
SUV and 1p/19q deletion status | through study completion, an average of 1 year
  Correlation between SUV and 1p/19q deletion status

CONTACTS AND LOCATIONS:
Overall Officials: Chen Xiao, Ph.D, Principal Investigator — Daping Hospital, Army Medical University
Locations (1):
- Department of Nuclear Medicine, Daping Hospital of Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jacobs SM, Wesseling P, de Keizer B, Tolboom N, Ververs FFT, Krijger GC, Westerman BA, Snijders TJ, Robe PA, van der Kolk AG. CXCR4 expression in glioblastoma tissue and the potential for PET imaging and treatment with [68Ga]Ga-Pentixafor /[177Lu]Lu-Pentixather. Eur J Nucl Med Mol Imaging. 2022 Jan;49(2):481-491. doi: 10.1007/s00259-021-05196-4. Epub 2021 Feb 7. PMID 33550492